CLINICAL TRIAL: NCT00501800
Title: Genetic Epidemiology of Ovarian Aging
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Aging (NIA) (NIH); Kaiser Foundation Research Institute (Other); Stanford University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: R01HD044876 (NIH); 5R01HD044876 (NIH)
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Infertility
Keywords: Reproductive Health; Fertility; Infertility; Genetics; Continental Population Groups; Epidemiology; Aging; Health
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Caucasian
- African American
- Chinese
- Latina (Mexican or Central American)
- Filipina

SUMMARY:
The purpose of this study is to identify clinical and genetic markers of ovarian aging. In this process, we will evaluate environmental factors that may affect fertility and the age at which fertility declines, and may influence the age at which women enter menopause. Wide variability exists between women both in the age at which menopause occurs and the rate of decline in oocyte number and reproductive capability. As the loss of ovarian function has profound impact on women's hormonal milieu and their subsequent risk for the development of disease, improving our understanding of the factors that determine the timing and rate of reproductive aging is critical to improving quality of life for all women. In addition, improving our understanding of reproductive aging has profound economic, and social, implications given the complex choices women face regarding the timing of childbearing and the growing burden of infertility. While the inter-individual variability in age at menopause has a large genetic component and possible environmental influences, to date no studies have addressed the relationship between oocyte number as reflected by antral follicle count (AFC) and genetic inheritance.

We hypothesize that ovarian aging, as reflected by antral follicle count, is largely determined by common genetic polymorphisms that impact the initial oocyte endowment and/or the rate of oocyte loss over time thus lowering antral follicle count for any given age. We further hypothesize that antral follicle count will be an improved marker of ovarian aging. Thus, we propose a study of the genetic and environmental factors that influence age-specific variability in antral follicle count.

DETAILED DESCRIPTION:
This is a cross-sectional study with a subgroup followed longitudinally over time. This study consists of four basic components:

* identification and recruitment of a population-based sample of 1,250 regularly cycling women of diverse ethnicities, ages 25-45;
* a baseline examination on days 2-4 of the menstrual cycle, including a blood draw, transvaginal ultrasound examination, body size measurements, and questionnaires, to establish cross-sectional relations between the AFC and the genetic and environmental exposures of interest (see Specific Aims);
* genetic analyses of X-chromosome and autosomal mutations, deletions, and polymorphisms, implicated in the control of ovarian function; and
* follow-up examination, 3 years after baseline, completed by approximately one-third of the cohort (n=450), to begin to describe longitudinal relations between AFC and the exposures of interest and to identify markers predictive of accelerated follicle loss.

Specific Aims:

1. Characterize antral follicle count (AFC) as a marker of ovarian age by comparing it to other available biomarkers, Follicle Stimulating Hormone (FSH), FSH/Lutenizing Hormone (LH), and inhibin B, and determine effect modification of these relationships by age.
2. Examine the relationship between antral follicle counts and the frequencies of specific genetic polymorphisms in the Deleted in AZoospermia-Like (DAZL) and interacting protein genes.
3. Determine the associations between race/ethnicity, body fat, and active and passive smoking and AFC, independently of age; if main effects are observed between genetic polymorphisms and AFC (Specific Aim 2), explore the effect modification of those relationships by race/ethnicity, body fat and active and passive smoking.
4. Determine the change in AFC over a three-year period and its relation to genetic and environmental characteristics, based on the approximately 450 women who complete a 3-year follow-up examination.

The primary goal of this study is to demonstrate the relationship between antral follicle count and common genetic polymorphisms and the effect of modification of environmental factors. To achieve this goal, our multidisciplinary team proposes to recruit a random sample of 1,250 regularly cycling, ethnically diverse women, ages 25-45, who belong to the Northern California Kaiser Permanente Medical Care (KPMC) Program in San Francisco.

This study will provide evidence to support ultrasound evaluation as a non-invasive marker of ovarian aging. This and the genetic testing may lead to an opportunity for prospective identification of patients at risk for early decline in ovarian function. The ability to accurately generate and share this type of information will allow women to become proactive in managing their fertility as well as to better understand their risks associated with reproductive aging. The recruitment of a large, population-based cohort will increase the generalizability of the data generated. The ethnic diversity of this population will allow multiple comparisons to identify true "risk factors" for early, and/or accelerated, ovarian aging and their correlation with ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-45 years
* Self-identifying as one of five specified race/ethnicities - Caucasian, Chinese, Filipino, African-American, or Hispanic (Mexican or Central American).
* Regular menstrual cycles (monthly bleeding with an interval of 25-35 days)
* Uterus and ovaries required.

Exclusion Criteria:

* Chronic medical illness such as heart, kidney, or liver disease or diabetes
* Endometriosis of ovary
* Prior surgical procedure for removal of ovarian cyst(s)
* Epilepsy
* Lupus
* Invasive cancer excluding squamous or basal cell skin cancers
* Prior treatment with chemotherapy or radiation therapy
* Use of any oral/systemic estrogen or progestin containing medication within a 3-month period
* Use of any central nervous system active medications known to disrupt the menstrual cycle (e.g. clonidine, aldomet)
* Psychiatric history involving functionally debilitating disturbance such as psychosis or major mood disorder requiring hospitalization or change in occupational or social functioning.
* Currently pregnant or breastfeeding
* Unable to speak and read English, Cantonese, or Spanish
* Concurrent participation in a clinical drug trial.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Population will be drawn from members of Northern California Kaiser Permanente Health Plan utilizing the Kaiser Permanente Division of Research database to identify potentially eligible subjects.
Sampling Method: Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2006-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Antral Follicle Counts | December 2014
  AFC as measured by Transvaginal Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle I. Cedars, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States